CLINICAL TRIAL: NCT01690832
Title: Fenoldopam for Prevention of Acute kidNey Injury in Patients With aCute coronarY Syndrome Undergoing Coronary Angiography and/or Percutaneous Coronary Intervention - The FANCY Trial
Brief Title: Fenoldopam for Prevention of Acute Kidney Injury
Acronym: FANCY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 595/2012/D
Record Dates: First submitted 2012-09-19; First posted 2012-09-24 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Coronary Artery Disease
Keywords: Contrast induced acute kidney injury
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard saline infusion (Active Comparator): standard i.v. 1 ml/kg/h saline infusion from 6 hours before the procedure to 12 hours after the procedure.
  Interventions: Drug: standard saline infusion
- fenoldopam infusion (Active Comparator): combination of i.v. 1 ml/kg/h saline infusion and fenoldopam administration (0.08 mcg/Kg/min) from 6 hours before the procedure to 12 hours after the procedure.
  Interventions: Drug: standard saline infusion; Drug: fenoldopam infusion

INTERVENTIONS:
Drug: standard saline infusion — i.v. 1 ml/kg/h saline infusion from 6 hours before the procedure to 12 hours after the procedure
  Other Names: saline infusion
Drug: fenoldopam infusion — combination of i.v. 1 ml/kg/h saline infusion and fenoldopam administration (0.08 mcg/Kg/min) from 6 hours before the procedure to 12 hours after the procedure
  Other Names: fenoldopam administration (0.08 mcg/Kg/min)
  Arms: fenoldopam infusion

SUMMARY:
Patients with acute coronary syndromes (ACS) are at increased risk for acute kidney injury (AKI) when they undergo urgent/emergency coronary angiography.

The optimal medical treatment for preventing the occurrence of contrast induced - acute kidney injury is still controversial.

Fenoldopam mesylate is a dopamine A1 receptor agonist that augments renal plasma flow that has reduced the risk of radiocontrast dye nephropathy in some (but not all) preliminary studies.

Neutrophil gelatinase-associated lipocalin (NGAL) is a new biomarker predictive for AKI already shown to be useful for earlier diagnosis of contrast induced nephropathy.

The primary objective of this study is to to test the hypothesis that fenoldopam, in addition to standard treatment, reduce the occurrence of contrast induced - acute kidney injury in patients with acute coronary syndrome (ACS) undergoing urgent/emergency coronary angiography and/or percutaneous coronary intervention.

DETAILED DESCRIPTION:
Patients with acute coronary syndromes (ACS) are at increased risk for acute kidney injury (AKI) when they undergo urgent/emergency coronary angiography.

The optimal medical treatment for preventing the occurrence of contrast induced - acute kidney injury is still controversial.

Fenoldopam mesylate is a dopamine A1 receptor agonist that augments renal plasma flow that has reduced the risk of radiocontrast dye nephropathy in some (but not all) preliminary studies.

Neutrophil gelatinase-associated lipocalin (NGAL) is a new biomarker predictive for AKI already shown to be useful for earlier diagnosis of contrast induced nephropathy.

The primary objective of this study is to to test the hypothesis that fenoldopam, in addition to standard treatment, reduce the occurrence of contrast induced - acute kidney injury in patients with acute coronary syndrome (ACS) undergoing urgent/emergency coronary angiography and/or percutaneous coronary intervention.

Patients will be randomized to standard i.v. 1 ml/kg/h saline infusion (Gr. A, N= 50) or to a combination of i.v. 1 ml/kg/h saline infusion and fenoldopam administration (0.08 mcg/Kg/min) from 6 hours before the procedure to 12 hours after the procedure.

Primary End-points

• Incidence of contrast induced acute kidney injury

Secondary End-points

• Post-angiographic 48-h absolute increase in creatinine, absolute increase in estimated glomerular filtration rate, and Neutrophil gelatinase-associated lipocalin (NGAL) value

ELIGIBILITY:
Inclusion Criteria:

* Indication to urgent/emergency coronary angiography
* Normal renal function (eGFR> 60 ml/min/1.73 m2)
* Moderate or high Mehran's risk score for CIN (>11).
* Able to understand and willing to sign the informed CF

Exclusion Criteria:

• Women of child bearing potential patients must demonstrate a negative pregnancy test performed within 24 hours before CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Contrast induced acute kidney injury | 48 hour
  Incidence of contrast induced acute kidney injury at 48 hour post-procedural control

SECONDARY OUTCOMES:
Markers of kidney injury | 48 hour
  Post-angiographic 48-h absolute increase in creatinine, absolute increase in estimated glomerular filtration rate, and Neutrophil gelatinase-associated lipocalin (NGAL) value

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pelliccia, MD, Principal Investigator — Sapienza University
Locations (1):
- Sapienza University, Rome, Lazio, Italy

REFERENCES:
- [Derived] Esezobor CI, Bhatt GC, Effa EE, Hodson EM. Fenoldopam for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD012905. doi: 10.1002/14651858.CD012905.pub2. PMID 39607014